CLINICAL TRIAL: NCT03803605
Title: IGHID 11802 - Combination Therapy With the Novel Clearance Modality (VRC07-523LS) and the Latency Reversal Agent (Vorinostat) to Reduce the Frequency of Latent, Resting CD4+ T Cell Infection (The VOR-07 Study)
Brief Title: Study to Assess Safety and Activity of Combination Therapy of VRC07-523LS and Vorinostat on HIV-infected Persons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-1217; U01AI117844 (NIH)
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-07

CONDITIONS: HIV-1 Infection
Keywords: VRC07-523LS; Vorinostat; HIV-1; Suppressed; Latency; Reversal; Novel; Monoclonal; Agent; Antibody; Frequency; T Cell; Infection; ART; Resting
MeSH Terms: conditions — Infections | interventions — Vorinostat

STUDY DESIGN:
Intervention Model Description: Single Arm: All participants will receive combination therapy consisting of VRC07-523LS and Vorinostat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VRC07-523LS + Vorinostat (VOR) (Experimental): Participants will receive two series of combination therapy consisting of one (1) intravenous (IV) dose of VRC-HIVMAB075-00-AB (VRC07-523LS) followed by 10 oral (PO) doses of Vorinostat (VOR) taken every 72 hours.
  Interventions: Biological: VRC07-523LS; Drug: Vorinostat (VOR)

INTERVENTIONS:
Biological: VRC07-523LS — VRC07-523LS 40 mg/kg administered intravenously per series (total of 2 infusions administered)
  Other Names: VRC-HIVMAB075-00-AB
Drug: Vorinostat (VOR) — Vorinostat 400 mg administered orally every 72 hours for 10 doses per series (A total of 20 400-mg doses administered)
  Other Names: Zolinza

SUMMARY:
Adult participants (18-64 years old) with HIV-1 Infection on ART with a CD4 T cell count ≥ 350 cells/mm3 and viral suppression for ≥ 24 months will be enrolled on this study. Participants will receive two series of combination therapy consisting of one (1) intravenous (IV) dose of VRC-HIVMAB075-00-AB (VRC07-523LS) followed by 10 oral (PO) doses of Vorinostat (VOR) taken every 72 hours. Each series will last approximately 1 month and the two series will be separated by at least one month. Combination ART is maintained throughout the study. Participants will be on this study for approximately 28 weeks (or about 7 months).

The purpose of this study is to:

* Evaluate the safety of two series of a VRC07-523LS infusion followed by multiple oral doses of VOR
* Determine if combining VRC07-523LS and VOR can have an impact on non-active HIV virus.

DETAILED DESCRIPTION:
This is a phase I, single-site, open-label study to evaluate the effects of VOR given in combination with VRC07-523LS on persistent HIV-1 Infection in HIV-infected individuals suppressed on ART.

The investigators hypothesize that combination therapy with VRC07-523LS and VOR will be safe and well-tolerated by HIV-1-infected participants suppressed on ART.

In Step 1, all participants will undergo study screening and enrollment. Participants will complete a baseline Leukapheresis (#1). In order to advance to Step 2, participants must be found to have a baseline measurement of the frequency of resting CD4 T cell infection ≥ 0.3 infectious units per million (IUPM) determined by Quantitative Viral Outgrowth Assay (QVOA) (lower limit of detection is 0.03 IUPM), as a further decrease from this low frequency of infection cannot be definitively measured given the QVOA assay threshold.

These criteria assure that eligible enrolled participants will have a measurable endpoint, thus decreasing risk of study participation for participants who would not have a measurable outcome.

Participants progressing to Steps 2 and 3 will receive two series of a single VRC07-523LS infusion followed by multiple doses of VOR.

In the first series (Step 2), participants will receive one VRC07-523LS 40 mg/kg infusion (infusion #1) on Day 0 followed by the 1st dose of VOR 400 mg PO taken at home on Day 2. Participants will take VOR 400 mg PO every 72 hours for a total of 10 doses.

In the second series (Step 3), participants will receive one VRC07-523LS 40 mg/kg infusion (infusion #2) on Day 60 followed by the 1st (of the 2nd series of VOR) dose of VOR 400 mg PO on Day 62. As in the previous Step, participants will take VOR 400 mg PO every 72 hours for a total of 10 doses.

Step 4 consists of 2 visits. The post-study treatment leukapheresis (#2) will be completed 5 - 8 weeks after the 2nd VRC07-523LS infusion. The End of Study Visit (EOS) will be scheduled to 2 - 4 weeks following the final leukapheresis (#2) visit.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years and < 65 years of age
2. Ability and willingness of participant to give written informed consent. Note: Due to the lack of foreseeable benefit to study participants, mentally incompetent participants will not be enrolled.
3. HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral assay.

   A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
4. On continuous antiretroviral therapy (ART defined below under Inclusion Criterion #5) for at least 24 months prior to screening.

   Note: Continuous ART prior to screening is defined as not missing more than 9 total days in the 3 months prior to screening.
5. Permitted regimens include:

   1. At least 3 ART agents (not counting ritonavir if less than a 200 mg total daily dose or cobicistat as one of the agents)

      Note: One of the agents must include an integrase inhibitor, NNRTI (Non-Nucleoside Reverse Transcriptase Inhibitors), or a boosted-PI (protease inhibitor).

      OR
   2. Two ART agents in which one of the agents is either a boosted PI or an integrase inhibitor.

   Note: Other fully suppressive antiretroviral combinations will be considered on a case-by-case basis.

   Note: Prior changes in, or elimination of, medications for easier dosing schedule, intolerance, toxicity, improved side effect profile or within a drug class are permitted if an alternative suppressive regimen was maintained but not within 30 days prior to screening.

   Note: Changes in drug formulation or dose are allowed (e.g., tenofovir disoproxil fumarate (TDF) to tenofovir alafenamide (TAF), ritonavir to cobicistat, or separate ART agent dosing to fixed-dose combination), but none within 30 days prior to screening.
6. Ability and willingness of participant to continue ART throughout the study.
7. Able and willing to adhere to protocol therapy, schedule, and is judged adherent to antiretroviral therapy.
8. Plasma HIV-1 RNA <50 copies/mL at 3 time points in the previous 24 months prior to screening and never ≥50 copies/mL on 2 consecutive time points in the last 24 months.

   Note: The documented plasma HIV-1 RNA must be performed by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
9. At least 1 documented plasma HIV-1 RNA result <50 copies/mL ≥24 months but ≤ 36 months prior to screening.
10. Plasma HIV-1 RNA level <50 copies/mL on an FDA-approved HIV RNA assay at screening, performed at US CLIA Certified Laboratory (or its equivalent).
11. CD4 cell count ≥ 350 cells/mm³ obtained within 90 days prior to study entry, performed at any US CLIA Certified Laboratory (or its equivalent).
12. Hepatitis C (HCV) antibody negative result within 60 days prior to study entry or, if the participant is HCV antibody positive, a negative HCV RNA within 60 days prior to study entry .
13. Hepatitis B surface antigen (HBsAg) negative within 60 days prior to study entry.
14. Interferon-gamma release assay (IGRA) for tuberculosis (TB) with negative results within 60 days prior to study entry.

    Note: Participants with a prior positive TB IGRA and documented evidence of completed prophylaxis treatment may enroll in the study and do not need to undergo IGRA at screening. Participants with a prior positive IGRA who have not completed prophylaxis treatment will be excluded.
15. Men and women who are not of reproductive potential (see below) are eligible without requiring the use of contraceptives. Acceptable documentation of sterilization and menopause is specified below.

    a) Written or oral documentation communicated by clinician or clinician's staff of one of the following:
    1. Physician report/letter
    2. Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy in any partner assigned male sex at birth, hysterectomy, oophorectomy, non-surgical permanent sterilization, or tubal ligation.)
    3. Discharge summary
    4. Documented or participant-reported absence of a period for ≥ one year must be confirmed with Follicle stimulating hormone-release factor (FSH) measurement elevated into the menopausal range as established by the reporting laboratory.
16. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) while on study and for 4 months after their last infusion.
17. All men participating in sexual activity that could lead to pregnancy must agree to consistently use at least one of the following forms of birth control for at least 21 days prior to Visit 3 and for 4 months after their last infusion:

    a) Condoms (male or female) with or without a spermicidal agent b) Diaphragm or cervical cap with spermicide c) Intrauterine device (IUD) d) Tubal ligation e) Hormone-based contraceptive f) Successful vasectomy

    Note: For female partners who are receiving ritonavir or cobicistat, estrogen-based contraceptives are not reliable and an alternative method should be suggested.
18. Ability and willingness to provide adequate locator information.
19. Ability and willingness to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the protocol requirements.
20. Adequate vascular access for infusion and leukapheresis.
21. Able to swallow pills without difficulty.
22. Agrees not to enroll on another study of an investigational research agent during the study period.

    Note: Investigational research agent is defined as any unlicensed investigational drug not yet approved by the FDA for intended use in humans.
23. Adequate organ function as indicated by the following laboratory values:

Hematological: Absolute neutrophil count (ANC) ≥1,500 /mm^3; Platelets ≥125,000 / mm^3; Hemoglobin ≥ 13 g/dL (male) and ≥ 11 g/dL (females)

Coagulation: Prothrombin Time or International Normalized Ratio (INR) ≤1.5x upper limit of normal (ULN)

Chemistries: K+ levels - Within normal limits; Mg++ levels ≥ 1.2 milliequivalents/L but <1.5 x ULN; Glucose - Screening serum glucose ≤ Grade 1 (fasting or non- fasting); Albumin ≥ 3.3 g/dL

Renal: Creatinine clearance determined by the chronic kidney disease (CKD)-Epi equation

Hepatic: Serum total bilirubin - Total bilirubin < 1.5 X ULN. If total bilirubin is elevated, direct bilirubin must be < 2 times the ULN range.

Note: If participant is on an atazanavir-containing therapy, then a direct bilirubin should be measured instead of the total bilirubin and must be ≤ 1.0 mg/dL.; aspartate aminotransferase (AST, SGOT) and alanine transaminase (ALT, SGPT) ≤ 1.25 X ULN; Alkaline Phosphatase ≤ 2.0 X ULN; Lipase < 1.6 X ULN; Urinalysis: Urine Protein - Negative or trace allowed ULN = upper limit of normal

Exclusion Criteria:

1. Known allergy or sensitivity to components of VOR
2. Serious adverse reactions to VRC07-523LS formulation components, VRC01 or VRC01LS, including history of anaphylaxis and related symptoms such as hives, respiratory difficulties, angioedema, and/or abdominal pain.
3. Women without documentation of an FSH level indicating menopause, hysterectomy or bilateral oophorectomy, bilateral tubal ligation, or non-surgical sterilization.
4. Receipt of compounds with histone deacetylase (HDAC) inhibitor-like activity, such as valproic acid within 30 days prior to screening. Potential participants may screen after a 30-day washout period.
5. Any investigational research agent within 30 days before study entry.

   Note: Co-enrollment in observational only studies is permitted.

   Note: Co-enrollment in other studies using FDA approved medication that are not otherwise listed as prohibited will be evaluated by the study PI and permitted on a case by case basis.
6. Plasma HIV RNA ≥150 copies/mL in the 6 months prior to screening.
7. Weight > 115 kg
8. Untreated syphilis infection (defined as a positive rapid plasma reagin (RPR) without clear documentation of treatment).

   Note: In cases of untreated syphilis, participant may rescreen following documentation of adequate treatment of syphilis
9. Current treatment for HCV with antiviral therapy or participants who have received HCV treatment within 6 months prior to screening.
10. Use of any of the following within 90 days prior to entry: immunosuppressive, immunomodulatory, cytokine, or growth stimulating factors such as systemic corticosteroids, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, interferon (IFN), interleukin-2 (IL-2).

    Not Exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical steroids for mild, uncomplicated dermatitis; or [4] a single course of oral /parental prednisone or equivalent at doses <2mg/kg/day and length of therapy <11 days with completion at least 30 days prior to enrollment.
11. Current use of Coumadin, warfarin, or other Coumadin derivative anticoagulants.
12. Prior receipt of HIV immunotherapy within 6 months prior to screening.
13. Prior receipt of more than three doses of Vorinostat.
14. Prior receipt of humanized or human monoclonal antibodies (mAbs) within 2 months prior to screening, whether licensed or investigational, will have eligibility determined by the study PI on a case-by-case basis.
15. Received any infusion blood product, immune globulin, or hematopoietic growth factors within 90 days prior to study entry.
16. Pregnancy or breast-feeding.
17. History or other evidence of severe illness, malignancy, immunodeficiency other than HIV, or any other condition that would make the participant unsuitable for the study in the opinion of the investigator, for at least 90 days prior to screening.
18. History of autoimmune disease

    Not exclusionary: Persons with mild, stable, and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgement of the site investigator (or designee), is likely not subject to exacerbation and likely not to complicate adverse event (AE) assessments.
19. Use of topical steroids over a total area exceeding 15 cm-2 within 30 days prior to Screening.
20. Treatment for an active AIDS-defining opportunistic infection within 90 days prior to Screening.
21. History of malignancy within the last 5 years.

    Note: A history of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary with documentation of complete resection at least 3 months prior to enrollment).
22. Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease.
23. Known psychiatric, medical, occupational, or substance abuse disorders that would interfere with participant's ability to fully cooperate with the requirements of the trial as assessed by the study investigator (or designee).

    Specifically exclusionary: [1] recent psychosis; [2] ongoing risk for suicide; or [3] recent history of suicide attempt or gesture.
24. History or other clinical evidence of a significant medical condition that includes but is not limited to:

    a) A process that would affect the immune response b) A process that would require medication that affects the immune response c) Any contraindication to repeated injections, infusions, or blood draws d) A condition or process (e.g., chronic urticarial or recent injection or infusion with evidence of residual inflammation) for which signs and symptoms could be confused with reactions to the study product
25. Current anti-tuberculosis therapy
26. Diabetes Mellitus type 1

    Note: Individuals with type 2 diabetes who meet inclusion criteria for glucose (Inclusion Criterion #23) are not excluded.
27. History of coronary artery disease, congestive heart failure, or cardiac arrhythmia requiring current treatment prior to study screening.
28. Hypertension - Exclude for blood pressure consistently >150 mm Hg systolic and >100 mm Hg diastolic.

    Note: Elevated BP occurring during research leukapheresis procedures completed within the past 12 months are excluded from this requirement. Acceptable isolated elevations must be noted as acceptable and signed by study PI or designee.
29. Unstable asthma (e.g., sudden acute attacks occurring without an obvious trigger) or either of the following in the past 12 months:

    1. >1 exacerbation of symptoms treated with oral/parental corticosteroids;
    2. Emergency care, urgent care, hospitalization, or intubation for asthma.
30. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
31. Seizure disorder: History of seizure(s) within past three years or use of medications used to prevent or treat seizure(s) at any time within the past 3 years.
32. History of asplenia - absence of normal spleen function as indicated by:

    1. Splenectomy
    2. Sickle cell disease
33. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
34. Prisoner recruitment and participation is not permitted.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Gay, MD, MPH, Principal Investigator — UNC-Chapel Hill; David M Margolis, MD, Study Director — UNC-Chapel Hill
Locations (1):
- University of North Carolina Health Care, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gay CL, James KS, Tuyishime M, Falcinelli SD, Joseph SB, Moeser MJ, Allard B, Kirchherr JL, Clohosey M, Raines SLM, Montefiori DC, Shen X, Gorelick RJ, Gama L, McDermott AB, Koup RA, Mascola JR, Floris-Moore M, Kuruc JD, Ferrari G, Eron JJ, Archin NM, Margolis DM. Stable Latent HIV Infection and Low-level Viremia Despite Treatment With the Broadly Neutralizing Antibody VRC07-523LS and the Latency Reversal Agent Vorinostat. J Infect Dis. 2022 Mar 2;225(5):856-861. doi: 10.1093/infdis/jiab487. PMID 34562096
- [Derived] Day S, Mathews A, Blumberg M, Vu T, Rennie S, Tucker JD. Broadening community engagement in clinical research: Designing and assessing a pilot crowdsourcing project to obtain community feedback on an HIV clinical trial. Clin Trials. 2020 Jun;17(3):306-313. doi: 10.1177/1740774520902741. Epub 2020 Feb 3. PMID 32009466

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting the following advancement criteria in Step 1: a frequency of resting CD4+ T cell infection (RCI) >0.30 per million cells proceeded to Step 2 and received the study intervention.
Period: Overall Study
Arm/Group | VRC07-523LS + Vorinostat (VOR)
Started | 15
Step 1: Participants With an RCI Measurement > 0.30 Per Million Cells | 8
Steps 2-4: Participants Receiving Study Intervention | 8
Completed | 8
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | VRC07-523LS + Vorinostat (VOR)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 49 [26 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Grade 3 or Higher Treatment-Related Adverse Event (AE)
Description: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 was used to measure safety where Grade 3 is defined as severe and Grade 4 is defined as potentially life-threatening. Treatment-Related AEs assessments are considered related to study product as possible, probable, or definite as defined in the protocol.
Time Frame: First day of study treatment through end of study, a total of approximately 36 weeks
Measure: Number; unit: percentage of participants
Arm/Group | VRC07-523LS + Vorinostat (VOR)
Number analyzed (Participants) | 8
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: For all participants (n=15): from the signing of informed consent through completion of Baseline leukapheresis (Visit 2), approximately 10 weeks. For qualifying participants who advanced to Step 2 (n=8) and initiated treatment (Visit 3) through end of study (Visit 13) an additional 26 weeks. A combined overall total of 36 weeks for intervention-treated participants.
Description: Solicited adverse events were collected using diaries for 72 hours following each infusion of VRC07-523LS. For reactogenicity assessment, participants recorded local and systemic pre-defined adverse events. Unsolicited adverse events were actively assessed by study staff at each intervention.
Groups:
- All Enrolled Participants Completing Step 1 (Visits 1 and 2): Participants meeting enrollment criteria who completed a Baseline leukapheresis procedure.
- Participants Receiving VRC07-523LS + Vorinostat (VOR) (Step 2/Visits 3-13): Participants with a Baseline RCI > 0.30 per million cells who received two series of combination therapy consisting of one (1) intravenous (IV) dose of VRC-HIVMAB075-00-AB (VRC07-523LS) followed by 10 oral (PO) doses of Vorinostat (VOR) taken every 72 hours.
  VRC07-523LS: VRC07-523LS 40 mg/kg administered intravenously per series (total of 2 infusions administered)
  Vorinostat (VOR): Vorinostat 400 mg administered orally every 72 hours for 10 doses per series (A total of 20 400-mg doses administered)
Arm/Group | All Enrolled Participants Completing Step 1 (Visits 1 and 2) | Participants Receiving VRC07-523LS + Vorinostat (VOR) (Step 2/Visits 3-13)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 14/15 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Participants Completing Step 1 (Visits 1 and 2) (N=15) | Participants Receiving VRC07-523LS + Vorinostat (VOR) (Step 2/Visits 3-13) (N=8)
Procedural hypertension (Injury, poisoning and procedural complications) | 13 (14) | 7 (7) — During leukapheresis procedure
Tissue infiltration (General disorders) | 3 (4) | 0 (0) — During leukapheresis procedure
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) — During leukapheresis procedure
Vessel puncture site swelling (General disorders) | 1 (1) | 0 (0) — During leukapheresis procedure
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (4)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Blood HIV RNA increased (Investigations) | 0 (0) | 1 (1) — Viral load >50 copies/mL (160 copies/mL)
Blood pressure systolic increased (Investigations) | 0 (0) | 2 (2) — During infusion procedure
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (6)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03803605/Prot_SAP_000.pdf